CLINICAL TRIAL: NCT01011816
Title: A Multicenter, Randomized, Blinded, Saline-Controlled Trial of Resorbable Biologic Disc Augmentation for Treatment of Symptomatic Lumbar Internal Disc Disruption (IDD) With the Biostat® System
Brief Title: Treatment of Symptomatic Lumbar Internal Disc Disruption (IDD) With the Biostat® System
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Stopped prior to last subject's last extended follow-up visit (78 weeks) due to lack of efficacy at the primary study endpoint (26 weeks)
Sponsor: Spinal Restoration, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SR-BX01-2007
Record Dates: First submitted 2009-11-09; First posted 2009-11-11 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-05-16 (Estimated); Status verified 2014-05

CONDITIONS: Back Pain; Chronic Low Back Pain; Internal Disc Disruption; Degenerative Disc Disease
Keywords: intervertebral disk
MeSH Terms: conditions — Back Pain; Intervertebral Disc Degeneration | interventions — Fibrin Tissue Adhesive; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- BIOSTAT BIOLOGX (Experimental): One injection of up to 4 mL of BIOSTAT BIOLOGX Fibrin Sealant into a single lumbar intervertebral disc
  Interventions: Biological: BIOSTAT BIOLOGX
- Saline (Placebo Comparator): One injection of up to 4 mL of saline solution into a single lumbar intervertebral disc
  Interventions: Drug: Saline

INTERVENTIONS:
Biological: BIOSTAT BIOLOGX — One injection of up to 4 mL of BIOSTAT BIOLOGX Fibrin Sealant into a single lumbar intervertebral disc using the Biostat Delivery Device
  Other Names: Fibrin Sealant
  Arms: BIOSTAT BIOLOGX
Drug: Saline — One injection of up to 4 mL of saline using the Biostat Delivery Device
  Other Names: 0.9% w/v Sodium Chloride Injection, USP
  Arms: Saline

SUMMARY:
The purpose of this investigation is to establish the safety and efficacy of the Biostat System when used for treatment of chronic low back (lumbar) pain due to symptomatic internal disc disruptions (IDD) by comparing safety and efficacy outcome measures between one group receiving BIOSTAT BIOLOGX® Fibrin Sealant through the Biostat® Delivery Device and another group receiving a preservative-free normal saline control delivered with the Biostat Delivery Device.

DETAILED DESCRIPTION:
The Biostat System is a combination product combining a resorbable biologic product with a delivery device system used to prepare and insert the biologic material into a lumbar intervertebral disc.

Symptomatic IDD is defined as a painful disruption of the internal architecture of a lumbar intervertebral disc, which appears as fissures, cracks or tears within the internal structures of the disc. Pain arising from a lumbar disc may not only be perceived as pain located in the low back (axial pain) but also as somatic referred pain involving the posterior hips, buttocks, lateral hips, groin, or posterior thighs.

The diagnosis of symptomatic IDD cannot currently be made on the basis of imaging studies, physical examination, or symptoms alone, and is best established with meticulously conducted disc provocation studies (provocation discography) that include pressure manometry and identification of an adjacent normal disc.

This treatment and study are not designed for patients exhibiting other potential sources of chronic low back pain such as more advanced degenerative disc disease with significant loss of disc height (>33%), spinal stenosis, or spondylolisthesis (see Eligibility Criteria).

ELIGIBILITY:
Inclusion Criteria:

* Age 18 or older and skeletally mature.
* Voluntarily signs the subject informed consent form and agrees to the release of medical information for purposes of this study (HIPAA authorization).
* Physically and mentally able to comply with the protocol, including ability to read and complete required forms, and willing and able to adhere to the follow-up requirements of the protocol.
* Chronic low back pain for at least 6 months.
* Pretreatment baseline low back pain of at least 40 mm on a 100 mm visual analog scale.
* Pretreatment baseline Roland-Morris Disability Questionnaire score of at least 9 on the 24-point questionnaire.
* Leg pain, if present, is of nonradicular origin, i.e., not due to stimulation of nerve roots or dorsal root ganglion of a spinal nerve by compressive forces.
* Leg pain, if present, does not extend below the knee and is no greater than 50% of low back pain as measured on a visual analog scale. If bilateral leg pain, the worst leg pain is no greater than 50% of low back pain.
* Low back pain unresponsive to at least 3 months of nonoperative care, which may include bed rest, antiinflammatory and analgesic medications, chiropractic manipulations, acupuncture, massage, physical therapy or home-directed lumbar exercise program.
* Diagnostic medial branch block or facet joint injection between 18 months and 2 weeks prior to the study procedure indicates no facet joint involvement.
* Diagnosis of symptomatic lumbar (L1-L2 - L5-S1) internal disc disruption (IDD), which requires confirmation of discogenic pain at one or two contiguous levels through positive provocation discography performed between 18 months and 2 weeks prior to the study procedure using pressure manometry and identification of an adjacent nonpainful disc. The disc provocation studies must precisely demonstrate concordant pain (<50 psi above opening pressure) and must demonstrate a fissure(s) in the outer one-third of the posterior or lateral anulus.

Exclusion Criteria:

* Cauda equina syndrome.
* Active malignancy or tumor as source of symptoms.
* Current infection or prior history of spinal infection (e.g., discitis, septic arthritis, epidural abscess) or an active systemic infection.
* Previous lumbar spine surgery.
* Evidence of prior lumbar vertebral body fracture.
* Disc bulge/protrusion or focal herniation at the symptomatic level(s) > 4 mm.
* Presence of disc extrusion or sequestration.
* Leg pain is greater than 50% of low back pain as measured on a visual analog scale.
* Leg pain that extends below the knee.
* Lumbar intervertebral foramen stenosis at the affected level(s) resulting in significant spinal nerve root compression (effacement of the majority of periganglion fat and loss of CSF signal around the nerve rootlets).
* Symptomatic central vertebral canal stenosis or absolute sagittal vertebral canal diameter < 9mm.
* Loss of disc space height at the symptomatic level(s) greater than one-third of an adjacent normal disc (or of the expected height in the case of an L5-S1 disc).
* Spondylolisthesis (> Grade 1) with or without spondylolysis at the symptomatic level(s).
* Lumbar spondylitis or other undifferentiated spondyloarthropathy.
* Dynamic instability at the symptomatic level(s) on lumbar flexion-extension radiographs indicated by >4.5 mm of translation or angular motion >15° at L1-L2, L2-L3, or L3-L4; >20° at L4-L5; or >25° at L5-S1.
* Diagnostic medial branch block or facet joint injection indicate facet joint involvement.
* Diagnostic sacroiliac injection indicates sacroiliac joint involvement for those patients with pain in the sacral region.
* Sustained relief (>3 months) of low back pain obtained with epidural injection of corticosteroids.
* Symptomatic involvement of more than two lumbar disc levels determined from discography.
* Neurological examination shows findings of radiculopathy or a significant underlying neurological condition (motor strength <4; sensory assessment abnormal; or reflexes absent or hyperactive with clonus).
* Prior thermal intradiscal procedure (e.g., intradiscal electrothermal therapy, intradiscal radiofrequency thermocoagulation).
* Any lumbar intradiscal injection procedure other than discography (e.g., injection of corticosteroids, methylene blue, dextrose, or glucosamine and chondroitin sulfate).
* Significant systemic disease, including unstable angina, autoimmune disease, rheumatoid arthritis, and muscular dystrophy.
* Congenital or acquired coagulopathy or thrombocytopenia; or currently taking anticoagulant, antineoplastic, antiplatelet, or thrombocytopenia-inducing medications; or undergoing radiation therapy.
* History of unexplained, easy, or persistent bruising or bleeding, bleeding from the gums, or bleeding problems experienced in previous surgical procedures.
* Aspirin or aspirin-containing medication taken ≤ 7 days prior to the procedure.
* Known or suspected hypersensitivity or allergy to drugs or components of the fibrin sealant (fibrinogen, thrombin, aprotinin, CaCl2) used in the procedure.
* History of, or current psychiatric or psychological condition, or substance or alcohol abuse that would potentially interfere with the subject's participation in the study.
* Ongoing or previous participation in another drug or device clinical study within the previous 2 months.
* Subject known to be pregnant or nursing at time of enrollment or with plans to become pregnant within the planned length of follow-up.
* Body habitus precludes adequate fluoroscopic visualization for the procedure or the procedure is physically impossible using the device.
* Concomitant conditions requiring daily oral steroid use for more than 30 days in the preceding 90 days.
* Pending litigation against a health care professional, except where required by the insurer as a condition of coverage, personal injury compensation or litigation claims.
* Prisoner or active military personnel who would not be available for follow-up.
* Presence of ferromagnetic implants that would disallow MRI of the symptomatic disc(s).
* Active or pending workers' compensation claims.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2010-03; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin J Pauza, MD, Principal Investigator — Spine Specialists PA
Locations (20):
- United States (20):
  - Alabama Clinical Therapeutics, LLC, Birmingham, Alabama
  - HOPE Research Institute, Phoenix, Arizona
  - Pain Control Associates of San Diego, Chula Vista, California
  - Napa Pain Institute, Napa, California
  - California Spine Diagnostics, San Francisco, California
  - The Spine Institute, Santa Monica, California
  - The Pain Institute, Inc, Merritt Island, Florida
  - Millennium Pain Center, Bloomington, Illinois
  - The Spine Center, Baltimore, Maryland
  - Medical Advanced Pain Specialists Applied Research Center, Edina, Minnesota
  - NewSouth NeuroSpine Pain Center, Flowood, Mississippi
  - OrthoCarolina Spine Center, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - OrthoNeuro, Inc., New Albany, Ohio
  - Allegheny Pain Management, Altoona, Pennsylvania
  - Orthopaedic & Spine Specialists, York, Pennsylvania
  - Spine Specialists PA, Tyler, Texas
  - Virginia Spine Research Institute, Richmond, Virginia
  - Advanced Pain Management, Virginia Beach, Virginia
  - Bellingham Spine Pain Specialists PS, Bellingham, Washington

REFERENCES:
- [Background] Yin W, Pauza K, Olan WJ, Doerzbacher JF, Thorne KJ. Intradiscal injection of fibrin sealant for the treatment of symptomatic lumbar internal disc disruption: results of a prospective multicenter pilot study with 24-month follow-up. Pain Med. 2014 Jan;15(1):16-31. doi: 10.1111/pme.12249. Epub 2013 Oct 23. PMID 24152079
- [Background] Buser Z, Keulling F, Jane L, Liebenberg E, Tang J, Thorne K, Coughlin D, Lotz J. Fibrin injection stimulates early disc healing in the porcine model [NASS Abstract 199]. Spine Journal 9:105S, 2009.
- [Background] Buser Z, Kuelling F, Liu J, Liebenberg E, Thorne KJ, Coughlin D, Lotz JC. Biological and biomechanical effects of fibrin injection into porcine intervertebral discs. Spine (Phila Pa 1976). 2011 Aug 15;36(18):E1201-9. doi: 10.1097/BRS.0b013e31820566b2. PMID 21325992
- [Background] Pauza K, Yin W, Olan W, Doerzbacher JF. BIOSTAT BIOLOGX(R) intradiscal fibrin sealant used for treatment of chronic low back pain caused by lumbar disc disruption: results of a 12 month, prospective multicenter pilot study. Spine Arthroplasty Society Meeting, April 27-30, 2010; New Orleans, LA. Abstract 248.
- [Background] Yin W, Pauza K, Olan W, Doerzbacher JF. Long-term outcomes from a prospective, multicenter investigational device exemption (IDE) pilot study of intradiscal fibrin sealant for the treatment of discogenic pain [ISIS Abstract]. Pain Medicine 12:1446-1447, 2011
- [Background] Buser Z, Liu J, Thorne KJ, Coughlin D, Lotz JC. Inflammatory response of intervertebral disc cells is reduced by fibrin sealant scaffold in vitro. J Tissue Eng Regen Med. 2014 Jan;8(1):77-84. doi: 10.1002/term.1503. Epub 2012 May 18. PMID 22610998

RESULTS

PARTICIPANT FLOW:
Groups:
- Saline: One injection of up to 4 mL of saline solution into a single lumbar intervertebral disc using the Biostat Delivery Device
Period: 26-Week Primary Endpoint
Arm/Group | BIOSTAT BIOLOGX | Saline
Started | 164 | 56
Completed | 157 | 54
Not Completed | 7 | 2
Period: 78-Week Extended Follow-up
Arm/Group | BIOSTAT BIOLOGX | Saline
Started | 157 | 54
Completed | 85 | 26
Not Completed | 72 | 28

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BIOSTAT BIOLOGX | Saline | Total
Number analyzed (Participants) | 164 | 56 | 220
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.7 (10.7) | 41.9 (11.4) | 40.2 (10.9)
Age, Customized [Number; unit: participants]
  ≥18-≤29 years | 30 | 11 | 41
  ≥30-≤39 years | 50 | 12 | 62
  ≥40-≤49 years | 51 | 20 | 71
  ≥50-≤59 years | 28 | 9 | 37
  ≥60 years | 5 | 4 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 83 | 32 | 115
  Male | 81 | 24 | 105
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 5 | 13
  Not Hispanic or Latino | 156 | 51 | 207
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 15 | 2 | 17
  White | 147 | 52 | 199
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.0 (6.1) | 27.5 (5.6) | 27.9 (5.9)
Currently Employed [Number; unit: participants]
  Yes | 96 | 34 | 130
  No | 65 | 22 | 87
  No Response | 3 | 0 | 3
Smoking Status [Number; unit: participants]
  Never | 90 | 21 | 111
  Previous | 46 | 19 | 65
  Current | 28 | 16 | 44
Previous Back Surgery [Number; unit: participants]
  None | 161 | 55 | 216
  Cervical | 3 | 1 | 4
History Low Back Pain [Number; unit: participants]
  0.5 - 1 year | 7 | 3 | 10
  1 - <5 years | 76 | 24 | 100
  5 - <10 years | 41 | 9 | 50
  10 - <20 years | 32 | 12 | 44
  >=20 years | 8 | 8 | 16
History Right Leg Pain [Number; unit: participants]
  None | 118 | 40 | 158
  <1 year | 8 | 3 | 11
  1 - <2 years | 11 | 2 | 13
  2 - <3 years | 11 | 5 | 16
  3 - <4 years | 2 | 0 | 2
  >=4 years | 14 | 6 | 20
History Left Leg Pain [Number; unit: participants]
  None | 110 | 33 | 143
  <1 year | 11 | 6 | 17
  1 - <2 years | 7 | 2 | 9
  2 - <3 years | 14 | 7 | 21
  3 - <4 years | 3 | 1 | 4
  >=4years | 19 | 7 | 26
Baseline Opioid Medication for Back Pain [Number; unit: participants]
  Yes | 109 | 37 | 146
  No | 55 | 19 | 74
Lumbar Level Treated [Number; unit: participants]
  L3/L4 | 12 | 8 | 20
  L4/L5 | 48 | 11 | 59
  L5/S1 | 104 | 37 | 141
Reason for Stopping Injection [Number; unit: participants]
  Subject Discomfort | 4 | 2 | 6
  Maximum Pressure Reached | 91 | 6 | 97
  Total Available Volume Delivered | 68 | 45 | 113
  Other [investigator discretion; saline backflow] | 1 | 3 | 4
Maximum Injection Pressure [Mean (Standard Deviation); unit: psi] — n=163 BIOSTAT BIOLOGX n=55 Saline
  psi | 83.0 (29.3) | 49.7 (25.7) | 74.6 (31.9)
Injection Volume [Mean (Standard Deviation); unit: ml] | 2.8 (0.9) | 3.3 (0.8) | 2.9 (0.9)

OUTCOME MEASURES:

1. Primary Outcome: Subject Composite Success
Description: Subject success based on a composite of minimum 30% decrease in low back pain, 30% improvement in function, maintenance of neurological status, no secondary interventions, and no serious adverse events.
Time Frame: 26 weeks
Population: All subjects adjudicated as a success or failure. Missed 26-week visit counted as failure (7 BIOSTAT BIOLOGX; 2 Saline). Unblinded subjects counted as failures (2 BIOSTAT BIOLOGX).
Measure: Number; unit: percentage of subjects
Arm/Group | BIOSTAT BIOLOGX | Saline
Number analyzed (Participants) | 164 | 56
percentage of subjects | 33.5 | 39.3
Statistical Analysis 1: Comparison: BIOSTAT BIOLOGX vs Saline; Null: No differenc between the percent success of Saline and BIOSTAT BIOLOGX; Test type: Superiority or Other; p = 0.52, Fisher Exact

2. Secondary Outcome: Visual Analog Scale for Low Back Pain
Description: Percent of subjects achieving a minimum 30% decrease in pain from baseline.
  The visual analog scale is a horizontal 100 mm line anchored on the left with the words "No Pain" and on the right with the words "Worst Possible Pain". Scores were obtained by measuring the distance in millimeters from the left origin of the line (0) to the point indicated with a slash placed by the subject to indicate the subject's level of low back pain experienced over the last week.
Time Frame: 26-weeks
Population: All subjects assigned success or failure. Missed 26-week visit counted as failure (7 BIOSTAT BIOLOGX; 2 Saline). Unblinded subjects counted as failures (2 BIOSTAT BIOLOGX).
Measure: Number; unit: percentage of subjects
Arm/Group | BIOSTAT BIOLOGX | Saline
Number analyzed (Participants) | 164 | 56
percentage of subjects | 42.1 | 50.0

3. Secondary Outcome: Roland-Morris Disability Questionnaire Score
Description: Percent of subjects achieving a minimum 30% decrease in Roland-Morris Disability Questionnaire score
  The Roland-Morris Disability Questionnaire is a widely studied and frequently used instrument for the assessment of function and disability related to low back pain. The questionnaire consists of 24 statements related to how a subject's back condition affects various activities of daily living. Subjects marked whether the statement either applied to them or did not apply at the time they responded to the statements. The score is the total number of questions with which the subject agreed. A higher score indicates less function and greater disability.
Time Frame: 26-weeks
Population: All subjects assigned as success or failure. Missed 26-week visit counted as failure (7 BIOSTAT BIOLOGX; 2 Saline). Unblinded subjects counted as failures (2 BIOSTAT BIOLOGX).
Measure: Number; unit: percentage of subjects
Arm/Group | BIOSTAT BIOLOGX | Saline
Number analyzed (Participants) | 164 | 56
percentage of subjects | 52.4 | 50.0

ADVERSE EVENTS:
Time Frame: 78-weeks postprocedure or until study termination for those subjects not reaching the 78-week follow-up examination
Arm/Group | BIOSTAT BIOLOGX | Saline
Serious Adverse Events (participants affected / at risk) | 22/164 | 7/56
Other Adverse Events (participants affected / at risk) | 49/164 | 11/56
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOSTAT BIOLOGX (N=164) | Saline (N=56)
Myocardial Infarction (Cardiac disorders) | 1 (1) | 1 (1)
Adrenal Mass (Endocrine disorders) | 1 (1) | 0 (0)
Crohn's Disease (Gastrointestinal disorders) | 0 (0) | 1 (1)
Diverticular Perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Wrist Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 6 (7) | 1 (1)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Uterine Leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Cerebral Haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 0 (0)
Radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Completed Suicide (Psychiatric disorders) | 1 (1) | 0 (0)
Conversion Disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Eating Disorder (Psychiatric disorders) | 0 (0) | 1 (1)
Substance Abuse (Psychiatric disorders) | 0 (0) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 2 (2)
Uterine Haemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hysterectomy (Surgical and medical procedures) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BIOSTAT BIOLOGX (N=164) | Saline (N=56)
Back Pain (Musculoskeletal and connective tissue disorders) | 20 (21) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 13 (14) | 3 (3)
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 16 (16) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (7) | 2 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure restrictions:

* Sponsor can review results communication prior to public release and can embargo communications regarding trial results for up to 30 days from the time submitted for review.
* If the communication contains patentable invention information, disclosure may be delayed up to 6 months for patent application filing.
* If the communication contains confidential information, Sponsor will notify the PI to remove the confidential information prior to release.